CLINICAL TRIAL: NCT03423160
Title: A Novel Framework for Impaired Imitation in ASD
Status: Active, not recruiting | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Ericka Wodka, Clinical Director, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Other Study IDs: IRB00146732
Record Dates: First submitted 2018-01-24; First posted 2018-02-06 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Autism: Right-handed children, ages 8.0-12.9, diagnosed with high-functioning ASD (and no co-morbid conditions, excluding anxiety disorders)
  Interventions: Other: None--observational
- Control: Right-handed children, ages 8.0-12.9, with no neurological or psychiatric diagnoses, currently or by history
  Interventions: Other: None--observational

INTERVENTIONS:
Other: None--observational — Observational study of behavior and electrical brain activity

SUMMARY:
There is long-standing recognition that people with autism spectrum disorders (ASD) have difficulty imitating others' actions; some investigators have highlighted impaired imitation as being a core contributor to the development of autism. What is yet unknown is precisely how imitation in children with ASD differs from that of typically developing peers.The investigators have identified a task parameter that separates preserved from impaired gesture imitation in ASD: children with ASD have difficulty imitating when the task requires two separate movement elements be coordinated simultaneously. By contrast, imitation is relatively preserved when movement elements are performed serially. The coordination of simultaneous movements is a hallmark of actions performed in the real world. With an eye to optimizing common therapies that depend heavily on imitation, the next step is to tease apart where, in the chain from perception to action, the capacity limitation in simultaneous processing lies. This study will be conducted in about two days and will involve imitating gestures that are presented via video. In addition, an EEG will record the brain's electrical activity during certain tasks to assess how the brain responds when the imitation task is more or less difficult. Several other clinical and behavioral measures will also be used.

DETAILED DESCRIPTION:
Visuo-motor imitation (VMI) impairments are central to the pathogenesis and affect the treatment of autism spectrum disorders (ASD). Therapies most commonly used to enhance social, communicative, academic, adaptive and occupational function in individuals with ASD rely on imitation, and impairments in VMI represent a bottleneck to the efficiency and efficacy of these therapies. Furthermore, an influential psychological account suggests that imitation impairments lead to the development of the ASD phenotype. By studying precisely how VMI is impaired in ASD, it is possible both to enhance widespread therapies and possibly to alter the course of the disorder itself. Unfortunately, researchers currently know little about the precise nature of imitation impairments in ASD. Our laboratory has recently identified a promising specific task parameter that separates preserved from impaired gesture imitation in ASD: children with ASD have difficulty imitating when the task requires two separate movement elements be coordinated simultaneously. By contrast, imitation is relatively preserved when movement elements are performed serially. This finding has been subsequently validated in a published study and again replicated in preliminary data. Coordination of simultaneous movements is a hallmark of skills performed in the real world (shoe tying, eating with knife-and-fork, driving, communicating with simultaneous verbal and gestural language). In order to optimize common adaptive and social-communicative skill therapies, the next step is to tease apart where, in the chain from perception to action, the capacity limitation in simultaneous processing lies. To do this, the investigators propose a rigorous research plan that encompasses three complementary experimental approaches: systematic psychophysics, neuropsychological testing and EEG. The goal is to specifically dissect the contribution to the simultaneity bottleneck in perceptual vs. motor processes using psychophysical control experiments. Under the hypothesis that some children with ASD may have more perceptual limitations and others may have more motor limitations, the investigators will assess heterogeneity explicitly. It is then possible to relate perceptual and motor aspects of simultaneous gesture VMI to validated neuropsychological tests of known clinical attentional and perceptual deficits in ASD. Finally, in Aim 3, the investigators will directly interrogate visual and motor networks. EEG measures of task-related activation are sensitive to task load and can be differentially assessed in visual and motor networks. By assessing deficient event-related modulation of EEG activity in visual or motor networks to simultaneous (high-load) vs. serial (low-load) conditions, the investigators can pinpoint the bottleneck. In addition to providing an approach that is complementary to the behavioral measures of Aims 1 and 2, the results of the EEG study can pave the way for future biomarkers and neurostimulation therapies.

ELIGIBILITY:
General Inclusion Criteria:

Age 8 years, 0 months to 12 years, 11 months, 30 days

Informed consent is provided by a parent or guardian and assent is provided by the child

Wechsler Intelligence Scale for Children-IV (WISC-IV) Full Scale Intelligence Quotient (IQ) > than 80, unless there is a 12 point or greater index discrepancy, in which case either the Verbal Comprehension Index or Perceptual Reasoning Index must be > 80 and the lower of the two must be > 65

Right-handedness, based on the Physical and Neurological Examination for Subtle Signs (PANESS) and Edinburgh Handedness Inventory.

General Exclusion Criteria:

Presence or history of a definitive neurologic disorder including seizures (except for uncomplicated brief febrile seizures), tumor, severe head injury, stroke, lesion, history of skull surgery or disease (because it affects electroencephalogram [EEG] analysis) or history of significant EEG abnormality

Presence of a severe chronic medical disorder

Presence of a significant visual impairment (corrected vision at distance worse than 20/40)

History of alcohol/substance abuse or dependency

Excessive tactile sensitivity of the scalp

Contact sensitivity to skin care products or cosmetics (due to possibility for irritation from the EEG electrodes/paste)

Hair styles that would interfere with contact between the EEG cap and the scalp and cannot be removed

Chronic tics or other significant movement disorders

Pregnancy (because of potential and unknown effects on brain function with respect to the measures of this study).

Children will be excluded if they are in foster care. Parents may be the biological or adoptive parent as long as they are the child's legal guardian.

Parents of children in the study may not have a diagnosis of autism.

Additional eligibility criteria for each group are contained in the following sections:

Specific Inclusion/Exclusion Criteria for ASD Group:

Diagnosis of autism spectrum disorder (ASD) will be made conservatively using either the Autism Diagnostic Interview-Revised (ADI-R), or the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2). If circumstances dictate that an ADOS-2 cannot be administered, the Brief Observation of Symptoms of Autism (BOSA) will be administered in its place. The ADOS-2 or BOSA will be performed by a psychology associate trained in its administration and scoring. Children must meet diagnostic thresholds on these instruments, and the diagnosis will be confirmed using Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5), by a neurologist.

Children may not have a history of known etiology for autism (e.g., fragile X syndrome, Tuberous Sclerosis, phenylketonuria, congenital rubella) or history of documented prenatal/perinatal insult, and they will show no evidence of meeting criteria for additional psychiatric diagnoses including major depression, bipolar disorder, conduct disorder, or adjustment disorder, based on maternal and child responses from the Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children (K-SADS). Subjects with comorbid anxiety disorders, including generalized anxiety disorder, separation anxiety disorder, simple and social phobias, and obsessive-compulsive disorder (OCD), will be allowed to participate since anxiety is common in ASD, and similar repetitive repertoires resembling "obsessive-compulsive behavior" are components of the diagnostic criteria for ASD.

Children with a comorbid diagnosis of attention-deficit/hyperactivity disorder (ADHD) will also be included due to the frequent rates of comorbidity with ASD. Children on stimulant medication will have the medication held on the day of testing.

Specific Inclusion/Exclusion Criteria for Typically Developing (TD) Controls

Children will be included in the typically developing (TD) control group if they: (1) Do not meet published cutoff criteria for ASD on the Social Responsiveness Scale, second edition (SRS-2), (2) do not have a history of a developmental disorder or a psychiatric disorder based on maternal and child responses from the K-SADS (excluding simple or social phobia); and (3) are free of immediate family members (sibling, parent) with autism or other pervasive developmental disorder.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: See above
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychophysical measures of imitation | Day 1 or 2
  2-3 purpose-designed psychophysical measures of gesture imitation ability and its sub-components

SECONDARY OUTCOMES:
EEG measures of brain activity during gesture imitation | Day 1 or 2
  Event-related spectral perturbation associated with imitation task (and control tasks), at sites reflecting the activity of visuo-motor networks

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Ewen, MD, Principal Investigator — Hugo Moser Research Institute at Kennedy Krieger
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Submission of de-identified EEG data to the National Institutes of Mental Health Data Archive
Time Frame: As required